CLINICAL TRIAL: NCT02914522
Title: Combined Phase 2b/3, Double-Blind, Randomized, Placebo-Controlled Studies Evaluating the Efficacy and Safety of Filgotinib in the Induction and Maintenance of Remission in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Study to Evaluate the Efficacy and Safety of Filgotinib in the Induction and Maintenance of Remission in Adults With Moderately to Severely Active Ulcerative Colitis
Acronym: SELECTION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-418-3898; 2016-001392-78 (EudraCT Number)
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Induction Study (Cohort A): Filgotinib 200 mg (Experimental): Participants in Cohort A (biologic-naive) received filgotinib 200 milligrams (mg) and placebo-to-match (PTM) filgotinib 100 mg orally once daily for 10 weeks.
  Interventions: Drug: Filgotinib; Drug: PTM filgotinib
- Induction Study (Cohort A): Filgotinib 100 mg (Experimental): Participants in Cohort A (biologic-naive) received filgotinib 100 mg and PTM filgotinib 200 mg orally once daily for 10 weeks.
  Interventions: Drug: Filgotinib; Drug: PTM filgotinib
- Induction Study (Cohort A): Placebo (Placebo Comparator): Participants in Cohort A (biologic-naive) received PTM filgotinib 200 mg and PTM filgotinib 100 mg orally once daily for 10 weeks.
  Interventions: Drug: PTM filgotinib
- Induction Study (Cohort B): Filgotinib 200 mg (Experimental): Participants in Cohort B (biologic-experienced) received filgotinib 200 mg and PTM filgotinib 100 mg orally once daily for 10 weeks.
  Interventions: Drug: Filgotinib; Drug: PTM filgotinib
- Induction Study (Cohort B): Filgotinib 100 mg (Experimental): Participants in Cohort B (biologic-experienced) received filgotinib 100 mg and PTM filgotinib 200 mg orally once daily for 10 weeks.
  Interventions: Drug: Filgotinib; Drug: PTM filgotinib
- Induction Study (Cohort B): Placebo (Placebo Comparator): Participants in Cohort B (biologic-experienced) received PTM filgotinib 200 mg and PTM filgotinib 100 mg orally once daily for 10 weeks.
  Interventions: Drug: PTM filgotinib
- Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg (Experimental): Participants in the Filgotinib 200 mg arm who completed the Induction Study and achieved either Endoscopy/Bleeding/Stool Frequency (EBS) remission or Mayo Clinic Score (MCS) response at Week 10 were re-randomized at Week 11 into the Maintenance Study to receive filgotinib 200 mg and PTM filgotinib 100 mg for an additional 47 weeks (up to Week 58).
  Interventions: Drug: Filgotinib; Drug: PTM filgotinib
- Maintenance Study: Placebo From Induction Filgotinib 200 mg (Placebo Comparator): Participants in the Filgotinib 200 mg arm who completed the Induction Study and achieved either EBS remission or MCS response at Week 10 were re-randomized at Week 11 into the Maintenance Study to receive PTM filgotinib orally once daily for an additional 47 weeks (up to Week 58).
  Interventions: Drug: PTM filgotinib
- Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg (Experimental): Participants in the Filgotinib 100 mg arm who completed the Induction Study and achieved either EBS remission or MCS response at Week 10 were re-randomized at Week 11 into the Maintenance Study to receive filgotinib 100 mg and PTM filgotinib 200 mg for an additional 47 weeks (up to Week 58).
  Interventions: Drug: Filgotinib; Drug: PTM filgotinib
- Maintenance Study: Placebo From Induction Filgotinib 100 mg (Placebo Comparator): Participants in the Filgotinib 100 mg arm who completed the Induction Study and achieved either EBS remission or MCS response at Week 10 were rerandomized at Week 11 into the Maintenance Study to receive PTM filgotinib orally once daily for an additional 47 weeks (up to Week 58).
  Interventions: Drug: PTM filgotinib
- Maintenance Study: Placebo From Induction Placebo (Placebo Comparator): Participants in the Placebo arm who completed the Induction Study and achieved either EBS remission or MCS response at Week 10 were re-randomized at Week 11 into the Maintenance Study to receive PTM filgotinib for an additional 47 weeks (up to Week 58).
  Interventions: Drug: PTM filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablet(s) administered orally once daily
  Other Names: GS-6034; GLPG0634
  Arms: Induction Study (Cohort A): Filgotinib 100 mg; Induction Study (Cohort A): Filgotinib 200 mg; Induction Study (Cohort B): Filgotinib 100 mg; Induction Study (Cohort B): Filgotinib 200 mg; Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg; Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg
Drug: PTM filgotinib — Tablet(s) administered orally once daily

SUMMARY:
The primary objectives of this study are to evaluate the efficacy of filgotinib in the induction and maintenance treatment of moderately to severely active ulcerative colitis (UC) in participants who are biologic-naive and biologic-experienced.

Participants who complete the study, or met protocol specified efficacy discontinuation criteria will have the option to enter a separate, long-term extension (LTE) study (Gilead Study GS-US-418-3899: NCT02914535).

ELIGIBILITY:
Key Inclusion Criteria:

* Males or non-pregnant, non-lactating females, ages 18 to 75 years, inclusive based on the date of the screening visit
* Documented diagnosis of UC of at least 6 months AND with a minimum disease extent of 15 cm from the anal verge. Documentation should include endoscopic and histopathologic evidence of UC.
* A surveillance colonoscopy is required at screening in individuals with a history of UC for 8 or more years, if one was not performed in the prior 24 months
* Moderately to severely active UC
* Previously demonstrated an inadequate clinical response, loss of response to, or intolerance to at least 1 of the following agents (depending on current country treatment recommendations/guidelines): corticosteroids, immunomodulators, tumor necrosis factor alpha (TNFa) antagonists, or vedolizumab

Key Exclusion Criteria:

* Presence of Crohn's disease, indeterminate colitis, ischemic colitis, fulminant colitis, ulcerative proctitis, or toxic mega-colon
* Active tuberculosis (TB) or history of latent TB that has not been treated
* Use of any concomitant prohibited medications as described in the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1351 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (343):
- United States (61):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - VA Long Beach Healthcare System, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - South Denver Gastroenterology, PC, Lone Tree, Colorado
  - Connecticut GI PC-Research Division, Farmington, Connecticut
  - UF Health at Shands Hospital, Gainesville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Tampa General Hospital, Tampa, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Atlanta Gastroenterology Specialist, PC, Suwanee, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Clinical Trials Unit, Louisville, Kentucky
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Massachusetts General Hospital - Crohn's and Colitis Center, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Research Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NY Scientific, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Carolina's GI Research, LLC, Raleigh, North Carolina
  - Fargo Gastroenterology and Hepatology Clinic, Fargo, North Dakota
  - Consultants for Clinical Research, Cincinnati, Ohio
  - UC Health Physicians Clifton, Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
  - Rapid City Medical Center, Rapid City, South Dakota
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Vanderbilt University Medical Center - IBD Clinic, Nashville, Tennessee
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - DHAT Research Institute, Garland, Texas
  - Baylor College of Medicine- Baylor Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC, San Antonio, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Texas Digestive Disease Consultants, San Marcos, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Spring Gastroenterology, The Woodlands, Texas
  - HP Clinical Research, Bountiful, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Gastroenterology Associates Of Tidewater, Chesapeake, Virginia
  - Emeritas Research Group LLC, Lansdowne Town Center, Virginia
  - McGuire DVAMC, Richmond, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin
- Argentina (2):
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Instituto Médico Cer, Quilmes
- Australia (11):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Coastal Digestive Health, Mountain Creek, Queensland
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Austria (2):
  - Universitatsklinik Innsbruck, Innsbruck
  - AKH-Medizinische Universitat Wien, Vienna
- Belgium (4):
  - GZA Ziekenhuizen campus Sint-Vincentius, Antwerp
  - CUB Hopital Erasme, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Chretien (CHC) - Clinique Saint-Joseph, Liège
- Bulgaria (3):
  - MHAT Sveti Pantaleymon - Pleven OOD, Pleven
  - "MDHAT Dr. St.Cherkezov" AD, Veliko Tarnovo
  - MHAT "Sveta Petka" AD, Vidin
- Canada (5):
  - University of Calgary, Heritage Medical Research Clinic, Calgary, Alberta
  - The Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Hamilton Health Sciences Corporation, McMaster University Medical Centre, Hamilton, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Toronto Digestive Disease Associates Inc., Vaughan
- Croatia (2):
  - Clinical Hospital Dubrava, Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (4):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Oblastni nemocnice Mlada Boleslav, a.s., nemocnice Stredoceskeho kraje, Gastroenterologicke oddeleni, Mladá Boleslav
  - G.E.P. Clinic, s r.o., Prague
  - ISCARE a.s. (Klinicke centrum ISCARE), Klinicke a vyzkumne centrum pro strevni zanety, Prague
- France (19):
  - CHU Amiens Picardie, Amiens
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand - Hopital d'Estaing, Clermont-Ferrand
  - APHP - Hopital Beaujon - Clichy - Universite Paris VII, Clichy
  - CHU de Dijon Bourgogne - Hopital Francois Mitterand, Dijon
  - CHU Grenoble Alpes, La Tronche
  - Hopital Universitaire de Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Hopital Nord, Marseille
  - CHU de Montpellier-Hopital Saint Eloi, Montpellier
  - CHU Hotel-Dieu, Nantes
  - Hopital de l'Archet 2, Nice
  - Institut Mutualiste Montsouris, Paris
  - CHU de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - CHU de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - CHU de Nancy - Hopital Brabois Adultes, Vandœuvre-lès-Nancy
- Georgia (3):
  - Unimed Ajara LLC - Batumi Referral Hospital, Batumi
  - Medi Club Georgia LLC, Tbilisi
  - Ltd. Unimed Kakheti - Telavi Referral Hospital, Telavi
- Germany (18):
  - Charite Universitatsmedizin Berlin, Berlin
  - Charite - Universitatsmedizin Berlin, Berlin
  - DRK Kliniken Berlin - Westend - Klinik fuer Innere Medizin, Berlin
  - Stadtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitaetsklinik Koln, Cologne
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Westklinikum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hannover
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - Universitatsklinikum Jena, Jena
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - EUGASTRO GmbH, Leipzig
  - Klinikum Luneburg, Lüneburg
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Klinikum der Universitat Munchen - Grosshadern, München
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitatsklinikum Ulm, Zentrum Fur Innere Medizin, Ulm
- Greece (2):
  - General Hospital of Athens "Hippokratio", 2nd Internal Medicine Clinic of Athens University, Hepato-gastroenterology Unit, Athens
  - General Hospital of Nikaias "Agios Pentelleimon", Gastroenterology Department, Athens
- Hong Kong (3):
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Department of Medicine & Therapeutics, The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin
- Hungary (6):
  - Bekes Megyei Kosponti Korhaz, Dr. Rethy Pal Tagkorhaz, IV. Belgyogyaszat - 2. Gasztroenterologia, Békéscsaba
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Kozponti Felnott Szakrendelo, Budapest
  - Szent Janos Korhaz es Eszak-budai Egitett Korhazak, I. Belgyogyaszati - Gasztroenterologiai Osztaly, Budapest
  - Debreceni Egyetem Klinikai Kozpont, II. sz. Belgyogyaszati Klinika, Gasztroenterologia, Debrecen
  - Bugat Pal Korhaz, Belgyogyaszat, Gyöngyös
  - Karolina Korhaz es Rendelointezet, Altalanos Belgyogyaszat-Gasztroenterologia, Mosonmagyaróvár
- India (24):
  - Kaizen Hospital, Ahmedabad
  - M S Ramaiah Medical College and Hospital, Bangalore
  - Apollo Speciality Hospital, Chennai
  - VGM Hospital Institute of Gastroenterology, Coimbatore
  - Gleneagles Global Hospitals, Hyderabad
  - Citizens Specialty Hospital, Hyderabad
  - Centre for Liver Research & Diagnostics, Hyderabad
  - S.R.KallaMemorial Gastro.&General Hospital,, Jaipur
  - S.M.S Medical College & Hospitals, Jaipur
  - School of Digestive & Liver Diseases, Kolkata
  - Dayanand Medical College & Hospital, Ludhiana
  - Kasturba Medical College (KMC) Hospital, Mangaluru
  - Lokmanya Tilak Municipal General Hospital, Mumbai
  - Midas Multispeciality Hospital Pvt. Ltd, Nagpur
  - Suretech Hospital & Research Centre Ltd, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Grant Medical Foundation Ruby Hall Clinic, Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Gandhi Hospital, Secunderabad
  - Institute of Gastroenterology & Liver Disease, Sunshine Hospitals, Secunderabad
  - Surat Institute of Digestive Sciences, Surat
  - Kasturba Hospital Medical College, Udupi
  - Sterling Hospital, Vadodara
  - Samvedana Hospital, Varanasi
- Beaumont Hospital, Dublin, Ireland
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Italy (8):
  - UOC Gastroenterologia II, Castellana Grotte
  - U.O. Fisiopatologia Digestiva, Catanzaro
  - Ospedale Clinicizzato SS. Annunziata - Dipartimento di Medicina, Chieti
  - Endocsopia Digestiva Centralizzata - ASST Fatebenefratelli Sacco, Ospedale Fatebenefratelli e Oftalmico, Milan
  - UOC Gastroenterologia, Padua
  - Azienda Ospedaliero-Universitaria Pisana - Presidio Ospedaliero Cisanello, Pisa
  - UOC Gastroenterologia ed Endoscopia Digestiva, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (44):
  - Medical Hospital, Tokyo Medical and Dental University, Bunkyō City
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Hokkaido P.W.F.A.C Sapporo-Kosei General Hospital, Chūōku
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Tokai University Hachioji Hospital, Hachioji-shi
  - Hiroshima University Hospital, Hiroshima
  - Fukuoka University Hospital, Jonan-ku
  - Ofuna Chuo Hospital, Kamakura
  - Kitakyushu City Hospital Organization Kitakyushu Municipal Medical Center, Kitakyushu-shi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kurume University Hospital, Kurume-shi
  - Hidaka Coloproctology Clinic, Kurume-shi
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - The Jikei University Hospital, Minatoku
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka-shi
  - Iwate Medical University Hospital, Morioka
  - Aichi Medical University Hospital, Nagakute-shi
  - Nagasaki University Hospital, Nagasaki
  - Saiseikai Niigata Daini Hospital, Nishiku
  - Hyogo College of Medicine College Hospital, Nishinomiya
  - Okayama University Hospital, Okayama
  - Wakakusa-Daiichi Hospital, Osaka
  - Ishida IBD Clinic, Ōita
  - Kinshukai Infusion Clinic, Ōsaka
  - Osaka City University Hospital, Ōsaka
  - Shiga University of Medical Science Hospital, Ōtsu
  - Saga-Ken Medical Centre Koseikan, Saga
  - Saga University Hospital, Saga
  - Kitasato University Hospital, THE KITASATO INSTITUTE, Sagamihara
  - Tokito Clinic, Saitama
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Tokushukai Hospital, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - National Hospital Organization Sendai Medical Center, Sendai
  - Tokyo Yamate Medical Center, Shinjuku-ku
  - Osaka University Hospital, Suita
  - Kagawa Prefectural Central Hospital, Takamatsu
  - National Hospital Organization Takasaki General Medical Center, Takasaki-shi
  - Osaka Medical College Hospital, Takatsuki
  - Ieda Hospital, Toyota-shi
  - Wakayama Medical University Hospital, Wakayama
  - Colo-proctology Center Matsushima Clinic, Yokohama
  - Yokohama Health Medicine Association Kannai Suzuki Clinic, Yokohama
- Malaysia (3):
  - University Kebangsaan Malaysia Medical Centre, Cheras
  - Hospital Pulau Pinang, George Town
  - Hospital Queen Elizabeth, Kota Kinabalu
- PCR-Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli, Mexico
- Netherlands (3):
  - Academic Medical Center (AMC), Amsterdam
  - Gelre Hospital, Apeldoorn
  - University Medical Center Utrecht, Utrecht
- New Zealand (5):
  - Christchurch Hospital, Christchurch
  - Auckland City Hospital, Grafton
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Newtown
  - Bay of Plenty District Health Board - Tauranga Hospital, Tauranga
- Norway (2):
  - Vestre Viken Hospital Trust, Baerum Hospital, Drammen
  - Akerskus University Hospital, Lørenskog
- Poland (21):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Klinika Gastroenterologii i Chorob Wewnetrznych, Bialystok
  - VITAMED Galaj i Cichomski spolka jawna, Bydgoszcz
  - Gabinet Lekarski Janusz Rudzinski, Bydgoszcz
  - NZOZ INTER-MED, Centrum Endoskopowe, Częstochowa
  - Niepubliczny Zaklad Opieki Zdrowotnej ALL-MEDICUS, Katowice
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp.J., Ksawerów
  - Santa Familia, Centrum Badan, Profilaktyki i Leczenia, Lodz
  - Centrum Innowacyjnych Terapii Sp. z o.o., Piaseczno
  - Clinical Research Center Spolka z organiczna odpowiedzialnoscia Medic-R Sp. k., Poznan
  - Gabinet Lekarski Dr. Hab. N. Med. Bartosz Korczowski, Rzeszów
  - Endoskopia Sp. z o.o., Sopot
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - GASTROMED Kopon, Zmudzkinski i Wspolnicy Sp. j. Specjalistyczne Centrum Gastrologii i Endoskopii, Torun
  - H-T.Centrum Medyczne Spolka z Ograniczona Odpowiedzialnoscia Sp.K., Tychy
  - Centrum Zdrowia MDM, Warsaw
  - Bodyclinic, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administacji w Warszawie, Warsaw
  - Niepubliczny Zaklad Opieki Zrodotnej VIVAMED Jadwige Miecz, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (2):
  - Hospital da Senhora da Oliveira Guimaraes, E.P.E., Guimarães
  - Centro Hospitalar de Sao Joao, EPE, Porto
- Romania (4):
  - SC MedLife SA, Gastroenterologie, Bucharest
  - Spitalul Clinic Colentina - Sectia de Spitulal Clinic Colentina, Gastroenterologie, Bucharest
  - Cabinet Medical Individual Dr Tirnaveanue Amelita, Gastroenterologie, Oradea
  - Cabinet Particular Policlinic Algomed SRL, Timișoara
- Russia (15):
  - State Budgetary Healthcare Institution "Chelyabinski Regional Clinical Hospital", Chelyabinsk
  - State Budgetary Institution of Health Irkustsk Order "Badge of Honor" Regional Clinical Hospital, Irkutsk
  - Federal State Budgetary Institution of Science Federal Research Center of Nutrition, Biotechnology and Food Safety, Moscow
  - State Budgetary Healthcare Institution of Moscow "City Clinical Hospital # 24 of Healthcare Department of Moscow", Moscow
  - State Budgetary Healthcare Institution of Moscow Region "Moscow Regional Clinical Research Institute n.a. M.F. Vladimirskiy", Moscow
  - State Budgetary Healthcare Institution of Nizhny Novgorod Region "Nizhny Novgorod Regional Clinical Hospital n.a. N.A., Nizhny Novgorod
  - State Budgetary Institution of Health of Novosibirsk Region "City Clinical Hospital #12", Novosibirsk
  - State Budgetary Healthcare Institution of the Novosibirsk Region "State Novosibirsk Regional Clinical Hospital", Novosibirsk
  - Saint Petersburg State Budgetary Healthcare Institution "City Polyclinic #38", Saint Petersburg
  - "Riat" LLC, Saint Petersburg
  - "Scientific Research Centre ECO-safety" LLC, Saint Petersburg
  - "PolyClinic EXPERT" LLC, Saint Petersburg
  - State Healthcare Institution "Regional Clinical Hospital", Saratov
  - Treatment and Prevention Interdistrict Institution "Smolenskie kliniki" LLC, Smolensk
  - State Autonomous Health Institution of the Tyumen Region "Multidisciplinary Consultative and Diagnostic Center", Tyumen
- Zvezdara University Medical Center, Belgrade, Serbia
- Singapore General Hospital, Singapore, Singapore
- KM Management, s.r.o., Gastroenterologicke a hepatologicke centrum Nitra, Nitra, Slovakia
- South Africa (2):
  - Dr MJ Prins, Cape Town
  - Peermed Clinical Trial Centre, Johannesburg
- South Korea (9):
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Division of Gastroenterology, Department of Medicine, Samsung Medical Center, Seoul
  - Hyung Hee University Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (5):
  - Centro Medico Teknon, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (3):
  - Danderyds Sjukhus AB, Danderyd
  - Skane University Hospital, Malmo
  - Akademiska Sjukhuset, Uppsala
- Switzerland (2):
  - Gastroenterologische Praxis Balsiger, Seibold und Partner, Bern
  - Universitatsspital Zurich, Zurich
- Taiwan (4):
  - Changhua Christian Hospital, Chang-hua
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei, Taipei
  - Chang Gung Medical Foundation, Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District
- Ukraine (18):
  - Municipal Institution "Cherkasy Regional Hospital of Cherkasy Regional Council", Gastroenterology Department, Cherkasy
  - Municipal City Clinical Hospital of the Emergency Medical Care, 1 st Therapy Department. Danylo Halytsky Lviv National Medical, Chernivtsi
  - Regional Municipal Institution "Chernivtsi Regional Clinical Hospital", Surgical Department, Chernivtsi
  - State Institution "Institute of Gastroenterology of National Academy of Medical Sciences of Ukraine", Dnipropetrovsk
  - Ivanto-Frankivsk Central City Clinic Hospital, Therapy Department #1. State Higher Education Institution Ivano-Frankivsk National, Ivano-Frankivsk
  - Municipal Health Care Institution "Kharkiv City Clinical Hospital #2 named after prof. O. O. Shalimov", Proctology Department, Kharkiv
  - L.T. Mala State Institution "National Institute of Therapy of National Academy of Medical Sciences of Ukraine", Kharkiv
  - Municipal Institution of Health Care "Regional Hospital of War Veterans", Therapeutic Department No1, Kharkiv
  - Treatment and Diagnostic Center of Private Enterprise of Private Production Company "Acinus", Kropyvnytskyi
  - Kyiv City Clinical Hospital No. 18, Proctology Department, Kyiv
  - Municipal Non-profit Enterprise "Consultative and Diagnostic Center" of Pechersk District of Kyiv, Therapy Department, Kyiv
  - Odesa Clinical Railway Hospital Branch of "Healthcare Center" of Public joint stock company "Ukrainian Railway", Odesa
  - Municipal Institution "Odesa Regional Clinical Hospital", Regional Gastroenterology Center based on Surgery Department, Odesa
  - Ternopil University Hospital, Regional Center of Gastroenterology with Hepatology, Ternopil
  - Vinnytsia Regional Clinical Hospital of War Veterans, Therapy Department #1, Vinnytsia
  - M.I. Pyrogov Vinnytsia Regional Clinical Hospital, Gastroenterology Department, Vinnytsia
  - Medical Center LLC "Health Clinic", Vinnytsia
  - Municipal Institution "Zaporizhzhya Regional Clinical Hospital" of Zaporizhzhya Regional Council, Zaporizhzhya
- United Kingdom (13):
  - The Pennine Acute Hospitals NHS Trust, Bury
  - Cambridge University Hospital NHS Foundation Trust, Cambridge
  - Royal Derby Hospital, Derby
  - NHS Lothian, Edinburgh
  - Glasgow Clinical Research Facility - Queen Elizabeth University Hospital, Glasgow
  - NHS Greater Glasgow and Clyde, Glasgow
  - Wycombe Hospital, High Wycombe
  - Imperial College Healthcare NHS Trust, St Mary's Hospital, London
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich
  - Biomedical Research Unit, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - St Helens and Knowsley Teaching Hospitals NHS Trust, Prescot
  - Southampton National Institute for Health Research, Wellcome Trust Clinical Research Facility, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magro F, Rogler G, Feagan BG, Peyrin-Biroulet L, Oortwijn A, Cougnaud L, Faes M, Bauer Y, Randall M, Rudolph C, Reinisch W. Association between endo-histological outcomes and colonic mucosal transcriptomic profiles in patients with ulcerative colitis receiving filgotinib. J Crohns Colitis. 2026 Jan 22:jjaf228. doi: 10.1093/ecco-jcc/jjaf228. Online ahead of print. PMID 41569324
- [Derived] Nakase H, Danese S, Reinisch W, Ritter T, Liang Y, Wendt E, Levesque BG, Yoon OK, Tian Y, Zhuo L, Karouzakis E, Bauer Y, Oortwijn A, Kaise T, Malkov VA, Hibi T. Mediators of Filgotinib Treatment Effects in Ulcerative Colitis: Exploring Circulating Biomarkers in the Phase 2b/3 SELECTION Study. Inflamm Bowel Dis. 2025 Apr 10;31(4):1095-1108. doi: 10.1093/ibd/izae278. PMID 39656830
- [Derived] Schreiber S, Feagan BG, Louis E, Hisamatsu T, Hibi T, Dron L, Jamoul C, Patel H, Harris K, Taliadouros V, Oortwijn A, Peyrin-Biroulet L. Distinct trajectories of symptomatic response in ulcerative colitis during filgotinib therapy: A post hoc analysis from the SELECTION study. United European Gastroenterol J. 2024 Nov;12(9):1243-1255. doi: 10.1002/ueg2.12686. Epub 2024 Oct 25. PMID 39452892
- [Derived] Watanabe K, Peyrin-Biroulet L, Danese S, Fujitani Y, Faes M, Oortwijn A, Lindsay JO, Rogler G, Hibi T. Impact of Concomitant Thiopurine on the Efficacy and Safety of Filgotinib in Patients with Ulcerative Colitis: Post Hoc Analysis of the Phase 2b/3 SELECTION Study. J Crohns Colitis. 2024 Jun 3;18(6):801-811. doi: 10.1093/ecco-jcc/jjad201. PMID 38019901
- [Derived] Schreiber S, Rogler G, Watanabe M, Vermeire S, Maaser C, Danese S, Faes M, Van Hoek P, Hsieh J, Moerch U, Zhou Y, de Haas A, Rudolph C, Oortwijn A, Loftus EV Jr. Integrated safety analysis of filgotinib for ulcerative colitis: Results from SELECTION and SELECTIONLTE. Aliment Pharmacol Ther. 2023 Nov;58(9):874-887. doi: 10.1111/apt.17674. Epub 2023 Sep 18. PMID 37718932
- [Derived] Vermeire S, Feagan BG, Peyrin-Biroulet L, Oortwijn A, Faes M, de Haas A, Rogler G. Withdrawal and Re-treatment with Filgotinib in Ulcerative Colitis: Post Hoc Analyses of the Phase 2b/3 SELECTION and SELECTIONLTE Studies. J Crohns Colitis. 2024 Jan 27;18(1):54-64. doi: 10.1093/ecco-jcc/jjad123. PMID 37540206
- [Derived] Lu X, Zhou ZY, Xin Y, Wang MJ, Gray E, Jairath V, Lindsay JO. Matching-Adjusted Indirect Comparisons of Filgotinib vs Vedolizumab, Tofacitinib, and Ustekinumab for Moderately to Severely Active Ulcerative Colitis. Inflamm Bowel Dis. 2024 Jan 5;30(1):64-77. doi: 10.1093/ibd/izad037. PMID 36946138
- [Derived] Dotan I, Feagan BG, Taliadouros V, Oortwijn A, Rudolph C, de Haas A, Santermans E, Hsieh J, Peyrin-Biroulet L, Hibi T. Efficacy of Filgotinib in Patients with Ulcerative Colitis by Line of Therapy in the Phase 2b/3 SELECTION Trial. J Crohns Colitis. 2023 Aug 21;17(8):1207-1216. doi: 10.1093/ecco-jcc/jjad039. PMID 36928705
- [Derived] Schreiber S, Feagan BG, Peyrin-Biroulet L, Vermeire S, Faes M, Harris K, Oortwijn A, Daniele P, Patel H, Danese S. Filgotinib Improved Health-Related Quality of Life and Led to Comprehensive Disease Control in Individuals with Ulcerative Colitis: Data from the SELECTION Trial. J Crohns Colitis. 2023 Jun 16;17(6):863-875. doi: 10.1093/ecco-jcc/jjad018. PMID 36756874
- [Derived] Loftus EV, Vermeire S, Feagan BG, Le Brun FO, Oortwijn A, Moerch U, Sandborn WJ, Hibi T. Corticosteroid-Sparing Effects of Filgotinib in Moderately to Severely Active Ulcerative Colitis: Data from the Phase 2b/3 SELECTION Study. J Crohns Colitis. 2023 Mar 18;17(2):211-220. doi: 10.1093/ecco-jcc/jjac122. PMID 36006011
- [Derived] Feagan BG, Danese S, Loftus EV Jr, Vermeire S, Schreiber S, Ritter T, Fogel R, Mehta R, Nijhawan S, Kempinski R, Filip R, Hospodarskyy I, Seidler U, Seibold F, Beales ILP, Kim HJ, McNally J, Yun C, Zhao S, Liu X, Hsueh CH, Tasset C, Besuyen R, Watanabe M, Sandborn WJ, Rogler G, Hibi T, Peyrin-Biroulet L. Filgotinib as induction and maintenance therapy for ulcerative colitis (SELECTION): a phase 2b/3 double-blind, randomised, placebo-controlled trial. Lancet. 2021 Jun 19;397(10292):2372-2384. doi: 10.1016/S0140-6736(21)00666-8. Epub 2021 Jun 3. PMID 34090625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, New Zealand, North America, South America, Asia and Europe. The first participant was screened on 14 November 2016. The last study visit occurred on 31 March 2020.
Pre-assignment Details: 2040 participants were screened.
Groups:
- Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg: Participants in the Filgotinib 200 mg arm who completed the Induction Study and achieved either Endoscopy/Bleeding/Stool Frequency (EBS) remission or Mayo Clinic Score (MCS) response at Week 10 were re-randomized at Week 11 into the Maintenance Study to receive filgotinib 200 mg and PTM filgotinib 100 mg orally once daily for an additional 47 weeks (up to Week 58).
- Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg: Participants in the Filgotinib 100 mg arm who completed the Induction Study and achieved either EBS remission or MCS response at Week 10 were re-randomized at Week 11 into the Maintenance Study to receive filgotinib 100 mg and PTM filgotinib 200 mg orally once daily for an additional 47 weeks (up to Week 58).
- Maintenance Study: Placebo From Induction Placebo: Participants in the Placebo arm who completed the Induction Study and achieved either EBS remission or MCS response at Week 10 were re-randomized at Week 11 into the Maintenance Study to receive PTM filgotinib orally once daily for an additional 47 weeks (up to Week 58).
Period: Induction Study: Up to Week 11
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort A): Placebo | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg | Induction Study (Cohort B): Placebo | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Placebo
Started | 245 | 278 | 137 | 262 | 286 | 143 | 0 | 0 | 0 | 0 | 0
Completed | 235 | 256 | 127 | 234 | 262 | 127 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 22 | 10 | 28 | 24 | 16 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 6 | 4 | 18 | 14 | 10 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent | 4 | 11 | 4 | 6 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 1 | 3 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator's Discretion | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance With Study Drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not Receive Study Drug | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Study: Week 11 to Week 58
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort A): Placebo | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg | Induction Study (Cohort B): Placebo | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Placebo
Started | 0 (Participants achieved either EBS remission/MCS response at Week 10 continued into Maintenance Study.) | 0 (Participants achieved either EBS remission/MCS response at Week 10 continued into Maintenance Study.) | 0 (Participants achieved either EBS remission/MCS response at Week 10 continued into Maintenance Study.) | 0 | 0 | 0 (Participants achieved either EBS remission/MCS response at Week 10 continued into Maintenance Study.) | 202 (Participants achieved either EBS remission/MCS response at Week 10 continued into Maintenance Study.) | 99 (Participants achieved either EBS remission/MCS response at Week 10 continued into Maintenance Study.) | 179 (Participants achieved either EBS remission/MCS response at Week 10 continued into Maintenance Study.) | 91 (Participants achieved either EBS remission/MCS response at Week 10 continued into Maintenance Study.) | 93
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 150 | 41 | 104 | 42 | 64
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 52 | 58 | 75 | 49 | 29
Not completed — Protocol-specified Disease Worsening | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 49 | 53 | 39 | 21
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 10 | 4 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 3 | 0 | 1
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 6 | 3 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Investigator's Discretion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Non-compliance With Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set for the Induction Study (Cohorts A and B) included all participants who took at least 1 dose of study drug in the Induction Study.
Groups:
- Induction Study (Cohort A): Filgotinib 200 mg: Participants in Cohort A (biologic-naive) received filgotinib 200 mg and PTM filgotinib 100 mg orally once daily for 10 weeks.
- Total: Total of all reporting groups
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort A): Placebo | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg | Induction Study (Cohort B): Placebo | Total
Number analyzed (Participants) | 245 | 277 | 137 | 262 | 285 | 142 | 1348
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 234 | 261 | 129 | 243 | 264 | 128 | 1259
  >=65 years | 11 | 16 | 8 | 19 | 21 | 14 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 120 | 50 | 114 | 99 | 56 | 561
  Male | 123 | 157 | 87 | 148 | 186 | 86 | 787
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    Race: American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Race: Asian | 77 | 79 | 38 | 50 | 51 | 27 | 322
    Race: Black or African American | 2 | 3 | 1 | 4 | 6 | 3 | 19
    Race: White | 165 | 192 | 95 | 190 | 212 | 98 | 952
    Race: Other | 0 | 2 | 2 | 0 | 0 | 1 | 5
    Race: Not Permitted | 0 | 1 | 1 | 18 | 16 | 13 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    Ethnicity: Not Hispanic or Latino | 238 | 269 | 134 | 249 | 273 | 134 | 1297
    Ethnicity: Hispanic or Latino | 6 | 6 | 3 | 8 | 8 | 4 | 35
    Ethnicity: Not Permitted | 1 | 2 | 0 | 5 | 4 | 4 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 57 | 56 | 25 | 17 | 22 | 11 | 188
  United States | 14 | 33 | 19 | 36 | 58 | 21 | 181
  India | 55 | 49 | 27 | 8 | 3 | 3 | 145
  Japan | 15 | 16 | 6 | 29 | 29 | 14 | 109
  Ukraine | 33 | 46 | 24 | 1 | 2 | 0 | 106
  France | 1 | 1 | 1 | 32 | 26 | 19 | 80
  Germany | 1 | 3 | 0 | 31 | 26 | 9 | 70
  Russia | 21 | 10 | 12 | 6 | 9 | 1 | 59
  Italy | 4 | 6 | 1 | 15 | 19 | 12 | 57
  United Kingdom | 7 | 3 | 0 | 12 | 11 | 7 | 40
  Belgium | 0 | 0 | 0 | 16 | 14 | 6 | 36
  South Korea | 1 | 7 | 2 | 5 | 12 | 5 | 32
  Australia | 6 | 3 | 1 | 10 | 8 | 2 | 30
  Hungary | 9 | 8 | 3 | 0 | 5 | 2 | 27
  Romania | 3 | 3 | 2 | 3 | 5 | 3 | 19
  Switzerland | 0 | 0 | 0 | 7 | 5 | 7 | 19
  Canada | 2 | 2 | 1 | 3 | 5 | 4 | 17
  Czechia | 3 | 4 | 4 | 4 | 2 | 0 | 17
  Taiwan | 1 | 3 | 0 | 4 | 4 | 0 | 12
  Israel | 1 | 1 | 0 | 5 | 4 | 0 | 11
  New Zealand | 1 | 2 | 0 | 4 | 2 | 1 | 10
  South Africa | 0 | 3 | 2 | 2 | 1 | 0 | 8
  Spain | 0 | 1 | 0 | 1 | 4 | 2 | 8
  Austria | 0 | 0 | 0 | 3 | 2 | 2 | 7
  Croatia | 0 | 1 | 0 | 2 | 1 | 2 | 6
  Norway | 0 | 2 | 2 | 1 | 1 | 0 | 6
  Sweden | 0 | 0 | 1 | 1 | 1 | 3 | 6
  Bulgaria | 1 | 3 | 1 | 0 | 0 | 0 | 5
  Greece | 1 | 1 | 0 | 0 | 2 | 1 | 5
  Georgia | 1 | 2 | 1 | 0 | 0 | 0 | 4
  Hong Kong | 2 | 1 | 0 | 1 | 0 | 0 | 4
  Netherlands | 0 | 0 | 0 | 2 | 0 | 2 | 4
  Serbia | 1 | 2 | 1 | 0 | 0 | 0 | 4
  Slovakia | 2 | 0 | 0 | 0 | 0 | 2 | 4
  Argentina | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Malaysia | 0 | 2 | 1 | 0 | 0 | 0 | 3
  Ireland | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Portugal | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Mexico | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Singapore | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Induction Study: Percentage of Participants Who Achieved Endoscopy/Bleeding/Stool Frequency (EBS) Remission at Week 10
Description: EBS remission was defined as an endoscopic subscore of 0 or 1; rectal bleeding subscore of 0; and at least a 1-point decrease in stool frequency from baseline to achieve a subscore of 0 or 1. Endoscopic subscore range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease (spontaneous bleeding, ulceration); rectal bleeding subscore range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes; stool frequency subscore range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 stools more than normal. Total score for EBS ranged from 0 to 9 (sum of all subscores), with higher scores indicating more severe disease.
Time Frame: Week 10
Population: Full Analysis Set for the Induction study (Cohorts A and B) included all randomized participants who took at least 1 dose of study drug in the corresponding Induction study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort A): Placebo | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg | Induction Study (Cohort B): Placebo
Number analyzed (Participants) | 245 | 277 | 137 | 262 | 285 | 142
percentage of participants | 26.1 [20.4 to 31.8] | 19.1 [14.3 to 23.9] | 15.3 [8.9 to 21.7] | 11.5 [7.4 to 15.5] | 9.5 [5.9 to 13.0] | 4.2 [0.6 to 7.9]
Statistical Analysis 1: Comparison: Induction Study (Cohort A): Filgotinib 200 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p = 0.0157, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel(CMH) test was stratified by concomitant use of oral, systemic corticosteroids (Yes/No) and immunomodulators (Yes/No) at Day 1; Difference in Percentages = 10.8, 95% CI 2-sided [2.1 to 19.5]
Statistical Analysis 2: Comparison: Induction Study (Cohort A): Filgotinib 100 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p = 0.3379, Cochran-Mantel-Haenszel; CMH test was stratified by concomitant use of oral, systemic corticosteroids (Yes or No) and of immunomodulators (Yes or No) at Day 1; Difference in Percentages = 3.8, 95% CI 2-sided [-4.3 to 12.0]
Statistical Analysis 3: Comparison: Induction Study (Cohort B): Filgotinib 200 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.0103, Cochran-Mantel-Haenszel; CMH was stratified by concomitant use of corticosteroids and of immunomodulators at Day 1, and number of prior exposure to biologic agent (≤1,>1); Difference in Percentages = 7.2, 95% CI 2-sided [1.6 to 12.8]
Statistical Analysis 4: Comparison: Induction Study (Cohort B): Filgotinib 100 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.0645, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 3]; Difference in Percentages = 5.2, 95% CI 2-sided [-0.0 to 10.5]

2. Primary Outcome: Maintenance Study: Percentage of Participants Who Achieved EBS Remission at Week 58
Description: as for outcome 1
Time Frame: Week 58
Population: Full Analysis Set for the Maintenance Study included all participants randomized to either the filgotinib 200 mg or filgotinib 100 mg treatment groups in the Induction Study (Cohorts A and B) who achieved EBS remission or MCS response at Week 10, were rerandomized, and took at least 1 dose of study drug in the Maintenance Study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg: Participants in the Filgotinib 200 mg arm who completed the Induction Study and achieved either EBS remission or MCS response at Week 10 were re-randomized at Week 11 into the Maintenance Study to receive filgotinib 200 mg and PTM filgotinib 100 mg orally once daily for an additional 47 weeks (up to Week 58).
Arm/Group | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg
Number analyzed (Participants) | 199 | 98 | 172 | 89
percentage of participants | 37.2 [30.2 to 44.2] | 11.2 [4.5 to 18.0] | 23.8 [17.2 to 30.5] | 13.5 [5.8 to 21.1]
Statistical Analysis 1: Comparison: Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg vs Maintenance Study: Placebo From Induction Filgotinib 200 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; CMH test was stratified by concomitant use of corticosteroids and of immunomodulators at maintenance baseline; participation in Induction (A or B); Difference in Percentages = 26.0, 95% CI 2-sided [16.0 to 35.9]
Statistical Analysis 2: Comparison: Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg vs Maintenance Study: Placebo From Induction Filgotinib 100 mg; Test type: Superiority; p = 0.0420, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 10.4, 95% CI 2-sided [-0.0 to 20.7]

3. Secondary Outcome: Induction Study: Percentage of Participants Who Achieved MCS Remission at Week 10
Description: MCS remission was defined as having a MCS of 2 or less and no single subscore higher than 1. The MCS was composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 stools more than normal), and physician's global assessment (PGA). The PGA acknowledged the participant's daily recollection of abdominal discomfort and general sense of wellbeing, and other observations, such as physical findings and the participant's performance status. The PGA score ranged from 0 to 3 with higher score indicating the severe disease. Total score for MCS ranged from 0 to 12 (sum of all subscores), with higher scores indicating more severe disease.
Time Frame: Week 10
Population: Participants in the Full Analysis Set for the Induction Study (Cohorts A and B) were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort A): Placebo | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg | Induction Study (Cohort B): Placebo
Number analyzed (Participants) | 245 | 277 | 137 | 262 | 285 | 142
percentage of participants | 24.5 [18.9 to 30.1] | 17.0 [12.4 to 21.6] | 12.4 [6.5 to 18.3] | 9.5 [5.8 to 13.3] | 6.0 [3.0 to 8.9] | 4.2 [0.6 to 7.9]
Statistical Analysis 1: Comparison: Induction Study (Cohort A): Filgotinib 200 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p = 0.0053, Cochran-Mantel-Haenszel; CMH test is stratified by concomitant use of oral, systemic corticosteroids (Yes or No) and of immunomodulators (Yes or No) at Day 1; Difference in Percentages = 12.1, 95% CI 2-sided [3.8 to 20.4]
Statistical Analysis 2: Comparison: Induction Study (Cohort A): Filgotinib 100 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p = 0.2295, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Difference in Percentages = 4.6, 95% CI 2-sided [-3.1 to 12.2]
Statistical Analysis 3: Comparison: Induction Study (Cohort B): Filgotinib 200 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.0393, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 3]; Difference in Percentages = 5.3, 95% CI 2-sided [-0.1 to 10.7]
Statistical Analysis 4: Comparison: Induction Study (Cohort B): Filgotinib 100 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.5308, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 3]; Difference in Percentages = 1.7, 95% CI 2-sided [-3.1 to 6.6]

4. Secondary Outcome: Induction Study: Percentage of Participants Who Achieved an Endoscopic Subscore of 0 at Week 10
Description: Endoscopic subscore range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease (spontaneous bleeding, ulceration).
Time Frame: Week 10
Population: Participants in the Full Analysis Set for the Induction Study (Cohorts A and B) were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort A): Placebo | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg | Induction Study (Cohort B): Placebo
Number analyzed (Participants) | 245 | 277 | 137 | 262 | 285 | 142
percentage of participants | 12.2 [7.9 to 16.6] | 5.8 [2.8 to 8.7] | 3.6 [0.1 to 7.2] | 3.4 [1.0 to 5.8] | 2.1 [0.3 to 3.9] | 2.1 [0.0 to 4.8]
Statistical Analysis 1: Comparison: Induction Study (Cohort A): Filgotinib 200 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p = 0.0047, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Difference in Percentages = 8.6, 95% CI 2-sided [2.9 to 14.3]
Statistical Analysis 2: Comparison: Induction Study (Cohort A): Filgotinib 100 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p = 0.3495, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Difference in Percentages = 2.1, 95% CI 2-sided [-2.6 to 6.8]
Statistical Analysis 3: Comparison: Induction Study (Cohort B): Filgotinib 200 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.4269, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 3]; Difference in Percentages = 1.3, 95% CI 2-sided [-2.5 to 5.1]
Statistical Analysis 4: Comparison: Induction Study (Cohort B): Filgotinib 100 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.9987, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 3]; Difference in Percentages = -0.0, 95% CI 2-sided [-3.4 to 3.4]

5. Secondary Outcome: Induction Study: Percentage of Participants Who Achieved Geboes Histologic Remission at Week 10
Description: Geboes histologic remission was assessed using the Geboes histologic scores for evaluation of disease severity in ulcerative colitis and classifies histologic changes. Remission was defined as having Grade 0 of <= 0.3, Grade 1 of <= 1.1, Grade 2A of <= 2A.3, Grade 2B of 2B.0, Grade 3 of 3.0, Grade 4 of 4.0, and Grade 5 of 5.0. Possible scores are Grade 0: Architectural changes (0.0=No abnormality to 0.3=Severe diffuse or multifocal abnormalities); Grade 1: Chronic inflammatory infiltrate (1.0=No increase to 1.3=Marked increase); Grade 2A: Eosinophils in lamina propria (2A.0=No increase to 2A.3-=Marked increase; Grade 2B: Neutrophils in lamina propria (2B.0= No increase to 2B.3=Marked increase); Grade 3: Neutrophils in epithelium (3.0=None to 3.3=>50% crypts involved); Grade 4: Crypt destruction (4.0=none to 4.3=Unequivocal crypt destruction), and Grade 5: Erosions and ulcerations: (5.0=No erosion, ulceration or granulation to 5.4=Ulcer or granulation tissue).
Time Frame: Week 10
Population: Participants in the Full Analysis Set for the Induction study (Cohorts A and B) were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort A): Placebo | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg | Induction Study (Cohort B): Placebo
Number analyzed (Participants) | 245 | 277 | 137 | 262 | 285 | 142
percentage of participants | 35.1 [28.9 to 41.3] | 23.8 [18.6 to 29.0] | 16.1 [9.5 to 22.6] | 19.8 [14.8 to 24.9] | 13.7 [9.5 to 17.8] | 8.5 [3.5 to 13.4]
Statistical Analysis 1: Comparison: Induction Study (Cohort A): Filgotinib 200 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Difference in Percentages = 19.0, 95% CI 2-sided [9.9 to 28.2]
Statistical Analysis 2: Comparison: Induction Study (Cohort A): Filgotinib 100 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p = 0.0672, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Difference in Percentages = 7.8, 95% CI 2-sided [-0.7 to 16.2]
Statistical Analysis 3: Comparison: Induction Study (Cohort B): Filgotinib 200 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.0019, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 3]; Difference in Percentages = 11.4, 95% CI 2-sided [4.2 to 18.6]
Statistical Analysis 4: Comparison: Induction Study (Cohort B): Filgotinib 100 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.1286, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 3]; Difference in Percentages = 5.2, 95% CI 2-sided [-1.4 to 11.8]

6. Secondary Outcome: Induction Study: Percentage of Participants Who Achieved MCS Remission (Alternative Definition) at Week 10
Description: MCS remission (alternative definition) was defined as having rectal bleeding, stool frequency, and PGA subscores of 0 and an endoscopic subscore of 0 or 1; overall MCS of ≤ 1. MCS possible subscores: rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 stools more than normal), PGA subscore (range: 0 to 3 with higher score indicating the severe disease), and an endoscopic subscore (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]. Total score for MCS ranged from 0 to 12 (sum of all subscores), with higher scores indicating more severe disease.
Time Frame: Week 10
Population: Participants in the Full Analysis Set for the Induction Study (Cohorts A and B) were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort A): Placebo | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg | Induction Study (Cohort B): Placebo
Number analyzed (Participants) | 245 | 277 | 137 | 262 | 285 | 142
percentage of participants | 12.2 [7.9 to 16.6] | 8.7 [5.2 to 12.2] | 4.4 [0.6 to 8.2] | 3.8 [1.3 to 6.3] | 2.1 [0.3 to 3.9] | 2.1 [0.0 to 4.8]
Statistical Analysis 1: Comparison: Induction Study (Cohort A): Filgotinib 200 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p = 0.0105, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Difference in Percentages = 7.9, 95% CI 2-sided [1.9 to 13.8]
Statistical Analysis 2: Comparison: Induction Study (Cohort A): Filgotinib 100 mg vs Induction Study (Cohort A): Placebo; Test type: Superiority; p = 0.1062, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Difference in Percentages = 4.3, 95% CI 2-sided [-1.0 to 9.6]
Statistical Analysis 3: Comparison: Induction Study (Cohort B): Filgotinib 200 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.3084, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 3]; Difference in Percentages = 1.7, 95% CI 2-sided [-2.2 to 5.6]
Statistical Analysis 4: Comparison: Induction Study (Cohort B): Filgotinib 100 mg vs Induction Study (Cohort B): Placebo; Test type: Superiority; p = 0.9109, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 3]; Difference in Percentages = -0.0, 95% CI 2-sided [-3.4 to 3.4]

7. Secondary Outcome: Induction Study: Pharmacokinetic (PK) Parameter: Cmax of Filgotinib and Its Metabolite GS-829845
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: Predose and at 0.5, 1, 2, 3, 4 and 6 hours postdose at a single visit between Week 2 and Week 10
Population: PK Substudy Analysis Set included all randomized participants who took at least 1 dose of filgotinib, participated in the PK substudy, and had at least 1 nonmissing intensive concentration value for filgotinib and/or GS-829845 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg
Number analyzed (Participants) | 4 | 11 | 9 | 17
nanograms per milliliter (ng/mL)
  Filgotinib: number analyzed (Participants) | 4 | 10 | 9 | 17
  Filgotinib | 1746.3 (1244.05) | 725.1 (313.36) | 2283.3 (1012.03) | 977.9 (403.51)
  Metabolite GS-829845 | 3227.5 (1204.50) | 1812.2 (701.46) | 4373.3 (1121.58) | 2002.9 (598.73)

8. Secondary Outcome: Induction Study: PK Parameter: Tmax of Filgotinib and Its Metabolite GS-829845
Description: Tmax is defined as the time to reach maximum observed concentration of drug.
Time Frame: Predose and at 0.5, 1, 2, 3, 4 and 6 hours postdose at a single visit between Week 2 and Week 10
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg
Number analyzed (Participants) | 4 | 11 | 9 | 17
hour (h)
  Filgotinib: number analyzed (Participants) | 4 | 10 | 9 | 17
  Filgotinib | 1.50 [0.75 to 2.00] | 0.75 [0.50 to 3.00] | 1.00 [0.50 to 2.25] | 0.57 [0.42 to 3.00]
  Metabolite GS-829845 | 3.76 [2.00 to 4.00] | 3.00 [1.00 to 6.00] | 3.02 [2.13 to 6.00] | 3.00 [1.03 to 6.00]

9. Secondary Outcome: Induction Study: PK Parameter: AUCtau of Filgotinib and Its Metabolite GS-82984
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Predose and at 0.5, 1, 2, 3, 4 and 6 hours postdose at a single visit between Week 2 and Week 10
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hour*nanograms per milliliter (h*ng/mL)
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg
Number analyzed (Participants) | 4 | 11 | 9 | 17
hour*nanograms per milliliter (h*ng/mL)
  Filgotinib: number analyzed (Participants) | 4 | 10 | 8 | 15
  Filgotinib | 5501.3 (1956.39) | 1909.3 (788.13) | 6475.6 (1643.00) | 2492.3 (852.52)
  Metabolite GS-829845: number analyzed (Participants) | 4 | 10 | 7 | 15
  Metabolite GS-829845 | 57982.0 (17767.52) | 31187.9 (11858.78) | 80208.6 (25096.57) | 36075.6 (13396.86)

10. Secondary Outcome: Induction Study: PK Parameter: AUClast of Filgotinib and Its Metabolite GS-82984
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: Predose and at 0.5, 1, 2, 3, 4 and 6 hours postdose at a single visit between Week 2 and Week 10
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg
Number analyzed (Participants) | 4 | 11 | 9 | 17
h*ng/mL
  Filgotinib: number analyzed (Participants) | 4 | 10 | 9 | 17
  Filgotinib | 5537.3 (1900.93) | 1881.9 (797.51) | 6743.1 (1743.68) | 2420.3 (837.26)
  Metabolite GS-829845 | 60938.4 (6961.77) | 30643.2 (12935.37) | 79286.3 (27968.49) | 34385.6 (15160.15)

11. Secondary Outcome: Induction Study: PK Parameter: Ctau of Filgotinib and Its Metabolite GS-82984
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Predose and at 0.5, 1, 2, 3, 4 and 6 hours postdose at a single visit between Week 2 and Week 10
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg
Number analyzed (Participants) | 4 | 11 | 9 | 17
ng/mL
  Filgotinib: number analyzed (Participants) | 3 | 8 | 8 | 13
  Filgotinib | 12.0 (4.74) | 4.5 (3.61) | 36.6 (79.06) | 4.1 (3.05)
  Metabolite GS-829845: number analyzed (Participants) | 3 | 10 | 8 | 15
  Metabolite GS-829845 | 2050.0 (493.66) | 934.8 (372.68) | 2581.3 (777.07) | 1062.8 (463.67)

12. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved MCS Remission at Week 58
Description: MCS remission was defined as having a MCS of 2 or less and no single subscore higher than 1. The MCS was composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 stools more than normal), and PGA. The PGA acknowledged the participant's daily recollection of abdominal discomfort and general sense of wellbeing, and other observations, such as physical findings and the participant's performance status. The PGA score ranged from 0 to 3 with higher score indicating the severe disease. Total score for MCS ranged from 0 to 12 (sum of all subscores), with higher scores indicating more severe disease.
Time Frame: Week 58
Population: Participants in the Full Analysis Set for the Maintenance Study were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg: Participants in the Filgotinib 100 mg arm) who completed the Induction Study and achieved either EBS remission or MCS response at Week 10 were re-randomized at Week 11 into the Maintenance Study to receive filgotinib 100 mg and PTM filgotinib 200 mg orally once daily for an additional 47 weeks (up to Week 58).
Arm/Group | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg
Number analyzed (Participants) | 199 | 98 | 172 | 89
percentage of participants | 34.7 [27.8 to 41.5] | 9.2 [3.0 to 15.4] | 22.7 [16.1 to 29.2] | 13.5 [5.8 to 21.1]
Statistical Analysis 1: Comparison: Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg vs Maintenance Study: Placebo From Induction Filgotinib 200 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 25.5, 95% CI 2-sided [16.0 to 35.0]
Statistical Analysis 2: Comparison: Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg vs Maintenance Study: Placebo From Induction Filgotinib 100 mg; Test type: Superiority; p = 0.0658, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 9.2, 95% CI 2-sided [-1.1 to 19.5]

13. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved Sustained EBS Remission at Week 58
Description: Sustained EBS remission was defined as having achieved EBS remission at both Weeks 10 and 58.
Time Frame: Week 58
Population: Participants in the Full Analysis Set for the Maintenance Study were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg
Number analyzed (Participants) | 199 | 98 | 172 | 89
percentage of participants | 18.1 [12.5 to 23.7] | 5.1 [0.2 to 10.0] | 8.7 [4.2 to 13.2] | 7.9 [1.7 to 14.0]
Statistical Analysis 1: Comparison: Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg vs Maintenance Study: Placebo From Induction Filgotinib 200 mg; Test type: Superiority; p = 0.0024, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 13.0, 95% CI 2-sided [5.3 to 20.6]
Statistical Analysis 2: Comparison: Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg vs Maintenance Study: Placebo From Induction Filgotinib 100 mg; Test type: Superiority; p = 0.7951, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 0.9, 95% CI 2-sided [-7.0 to 8.7]

14. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved 6-Month Corticosteroid-Free EBS Remission at Week 58
Description: Six-month corticosteroid-free EBS remission at Week 58 was defined as achieving EBS remission with no corticosteroid use for the indication of ulcerative colitis for at least 6 months prior to Week 58.
Time Frame: Week 58
Population: Participants in the Full Analysis Set who were on corticosteroids at Maintenance Study baseline were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg
Number analyzed (Participants) | 92 | 47 | 81 | 37
percentage of participants | 27.2 [17.5 to 36.8] | 6.4 [0.0 to 14.4] | 13.6 [5.5 to 21.7] | 5.4 [0.0 to 14.0]
Statistical Analysis 1: Comparison: Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg vs Maintenance Study: Placebo From Induction Filgotinib 200 mg; Test type: Superiority; p = 0.0055, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 20.8, 95% CI 2-sided [7.7 to 33.9]
Statistical Analysis 2: Comparison: Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg vs Maintenance Study: Placebo From Induction Filgotinib 100 mg; Test type: Superiority; p = 0.1265, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 8.2, 95% CI 2-sided [-4.2 to 20.6]

15. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved Endoscopic Subscore of 0 at Weeks 58
Description: as for outcome 4
Time Frame: Week 58
Population: Participants in the Full Analysis Set for the Maintenance Study were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg
Number analyzed (Participants) | 199 | 98 | 172 | 89
percentage of participants | 15.6 [10.3 to 20.9] | 6.1 [0.9 to 11.4] | 13.4 [8.0 to 18.7] | 7.9 [1.7 to 14.0]
Statistical Analysis 1: Comparison: Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg vs Maintenance Study: Placebo From Induction Filgotinib 200 mg; Test type: Superiority; p = 0.0157, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 9.5, 95% CI 2-sided [1.8 to 17.1]
Statistical Analysis 2: Comparison: Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg vs Maintenance Study: Placebo From Induction Filgotinib 100 mg; Test type: Superiority; p = 0.1808, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 5.5, 95% CI 2-sided [-2.9 to 13.9]

16. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved Geboes Histologic Remission at Week 58
Description: as for outcome 5
Time Frame: Week 58
Population: Participants in the Full Analysis Set for the Maintenance Study were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg
Number analyzed (Participants) | 199 | 98 | 172 | 89
percentage of participants | 38.2 [31.2 to 45.2] | 13.3 [6.0 to 20.5] | 27.9 [20.9 to 34.9] | 18.0 [9.4 to 26.5]
Statistical Analysis 1: Comparison: Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg vs Maintenance Study: Placebo From Induction Filgotinib 200 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 24.9, 95% CI 2-sided [14.6 to 35.2]
Statistical Analysis 2: Comparison: Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg vs Maintenance Study: Placebo From Induction Filgotinib 100 mg; Test type: Superiority; p = 0.0521, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 9.9, 95% CI 2-sided [-1.3 to 21.2]

17. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved MCS Remission (Alternative Definition) at Week 58
Description: as for outcome 6
Time Frame: Week 58
Population: Participants in the Full Analysis Set for the Maintenance Study were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg
Number analyzed (Participants) | 199 | 98 | 172 | 89
percentage of participants | 22.1 [16.1 to 28.1] | 6.1 [0.9 to 11.4] | 12.2 [7.0 to 17.4] | 7.9 [1.7 to 14.0]
Statistical Analysis 1: Comparison: Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg vs Maintenance Study: Placebo From Induction Filgotinib 200 mg; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 16.0, 95% CI 2-sided [7.8 to 24.2]
Statistical Analysis 2: Comparison: Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg vs Maintenance Study: Placebo From Induction Filgotinib 100 mg; Test type: Superiority; p = 0.2946, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in Percentages = 4.3, 95% CI 2-sided [-3.9 to 12.6]

18. Secondary Outcome: Maintenance Study: Plasma Concentration of Filgotinib and Its Metabolite GS-829845
Description: Plasma concentration is defined as the measured drug concentration of filgotinib and its metabolite GS-829845. Lower limit of quantitation (LLOQ) was defined as 1 ng/mL for analyte filgotinib and 2 ng/mL for analyte GS-829845.
Time Frame: Week 26 (any Time) and Week 58 (predose)
Population: PK Analysis Set included all participants in the Safety Analysis Set who who took at least 1 dose of filgotinib and had at least 1 nonmissing plasma concentration value for filgotinib and/or its metabolite GS-829845 with available data were analyzed. Data was not collected for the Maintenance Study Placebo arms.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg
Number analyzed (Participants) | 173 | 136
ng/mL
  Filgotinib: Week 26: number analyzed (Participants) | 169 | 127
  Filgotinib: Week 26 | 8.5 [5.0 to 25.8] | 4.4 [2.5 to 14.0]
  Filgotinib: Week 58: number analyzed (Participants) | 44 | 26
  Filgotinib: Week 58 | 3.9 [NA to 9.1] — Value was below the limit of quantitation. | 4.1 [NA to 6.9] — Value was below the limit of quantitation.
  Metabolite GS-829845: Week 26: number analyzed (Participants) | 170 | 130
  Metabolite GS-829845: Week 26 | 2495.0 [1940.0 to 3010.0] | 1180.0 [852.0 to 1550.0]
  Metabolite GS-829845: Week 58: number analyzed (Participants) | 44 | 26
  Metabolite GS-829845: Week 58 | 1930.0 [1320.0 to 2630.0] | 973.5 [773.0 to 1350.0]

ADVERSE EVENTS:
Time Frame: Induction Study: first dose date up to one day before the Maintenance first dose date or last dose date whichever is earlier (maximum 17 weeks) plus 30 days, Maintenance study: First dose to the last dose in the Maintenance Study (maximum 51 weeks) plus 30 days
Description: Adverse Events: Safety Analysis Set for the study included all participants who took at least 1 dose of study drug in either the Induction Study (Cohorts A and B) or the Maintenance Study. All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized on Day 1 into each corresponding study.
Arm/Group | Induction Study (Cohort A): Filgotinib 200 mg | Induction Study (Cohort A): Filgotinib 100 mg | Induction Study (Cohort A): Placebo | Induction Study (Cohort B): Filgotinib 200 mg | Induction Study (Cohort B): Filgotinib 100 mg | Induction Study (Cohort B): Placebo | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg | Maintenance Study: Placebo From Induction Filgotinib 200 mg | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Filgotinib 100 mg | Maintenance Study: Placebo From Induction Placebo
All-Cause Mortality (participants affected / at risk) | 0/245 | 0/278 | 0/137 | 0/262 | 0/286 | 0/143 | 2/202 | 0/99 | 0/179 | 0/91 | 0/93
Serious Adverse Events (participants affected / at risk) | 3/245 | 13/277 | 4/137 | 19/262 | 15/285 | 9/142 | 9/202 | 0/99 | 8/179 | 7/91 | 4/93
Other Adverse Events (participants affected / at risk) | 40/245 | 43/277 | 20/137 | 83/262 | 77/285 | 55/142 | 67/202 | 33/99 | 53/179 | 33/91 | 26/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Study (Cohort A): Filgotinib 200 mg (N=245) | Induction Study (Cohort A): Filgotinib 100 mg (N=277) | Induction Study (Cohort A): Placebo (N=137) | Induction Study (Cohort B): Filgotinib 200 mg (N=262) | Induction Study (Cohort B): Filgotinib 100 mg (N=285) | Induction Study (Cohort B): Placebo (N=142) | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg (N=202) | Maintenance Study: Placebo From Induction Filgotinib 200 mg (N=99) | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg (N=179) | Maintenance Study: Placebo From Induction Filgotinib 100 mg (N=91) | Maintenance Study: Placebo From Induction Placebo (N=93)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 3 | 3 | 7 | 5 | 5 | 0 | 0 | 1 | 1 | 0
Dental cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Supernumerary teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Type I hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhagic infarction (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Study (Cohort A): Filgotinib 200 mg (N=245) | Induction Study (Cohort A): Filgotinib 100 mg (N=277) | Induction Study (Cohort A): Placebo (N=137) | Induction Study (Cohort B): Filgotinib 200 mg (N=262) | Induction Study (Cohort B): Filgotinib 100 mg (N=285) | Induction Study (Cohort B): Placebo (N=142) | Maintenance Study: Filgotinib 200 mg From Induction Filgotinib 200 mg (N=202) | Maintenance Study: Placebo From Induction Filgotinib 200 mg (N=99) | Maintenance Study: Filgotinib 100 mg From Induction Filgotinib 100 mg (N=179) | Maintenance Study: Placebo From Induction Filgotinib 100 mg (N=91) | Maintenance Study: Placebo From Induction Placebo (N=93)
Anaemia (Blood and lymphatic system disorders) | 6 | 10 | 4 | 12 | 11 | 10 | 4 | 0 | 4 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 3 | 8 | 7 | 9 | 8 | 6 | 6 | 2 | 4
Colitis ulcerative (Gastrointestinal disorders) | 6 | 3 | 5 | 14 | 11 | 6 | 21 | 18 | 18 | 16 | 10
Nausea (Gastrointestinal disorders) | 8 | 3 | 1 | 7 | 15 | 6 | 5 | 1 | 4 | 0 | 2
Pyrexia (General disorders) | 5 | 1 | 1 | 6 | 3 | 8 | 6 | 1 | 4 | 3 | 1
Nasopharyngitis (Infections and infestations) | 7 | 9 | 2 | 20 | 20 | 11 | 22 | 6 | 12 | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 13 | 4 | 5 | 11 | 3 | 6 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2 | 8 | 10 | 7 | 8 | 7 | 6 | 3 | 4
Headache (Nervous system disorders) | 11 | 12 | 6 | 19 | 10 | 9 | 7 | 0 | 10 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT02914522/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT02914522/SAP_001.pdf